CLINICAL TRIAL: NCT04687475
Title: Implementation of a Clinical Tool to Improve Waitlist Mortality in Patients With Cystic Fibrosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-112
Record Dates: First submitted 2020-12-17; First posted 2020-12-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis; Lung Transplant; Complications
MeSH Terms: conditions — Cystic Fibrosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Tool (Mobile Spirometry and Survey) (Experimental): All subjects enrolled will be placed into the clinical tool arm. The clinical tool is comprised of a mobile application based assessment of home spirometry and a survey measuring patient reported outcomes.
  Interventions: Other: Clinical Tool (Mobile Spirometry and Survey)

INTERVENTIONS:
Other: Clinical Tool (Mobile Spirometry and Survey) — The clinical tool is a combination of home spirometry measurements and a patient survey measuring patient reported outcomes including the Cystic Fibrosis Respiratory Symptom Diary (CFRSD) and Chronic Respiratory Infection Symptom Score (CRISS©), with permission from the Seattle Quality of Life Group.

SUMMARY:
Implementation of a Clinical Tool to Improve Waitlist Mortality in Patients With Cystic Fibrosis

DETAILED DESCRIPTION:
The aim of this project is to implement a clinical tool utilizing predictors of mortality for patients with Cystic Fibrosis (CF) on the waiting list to identify candidates that should present for urgent medical care and, if appropriate, will prompt clinicians to update a candidate's lung allocation score (LAS), the score used to prioritize lung transplant candidates for transplant by medical urgency, and avoid undetected decline. The clinical tool consists of home spirometry measures and patient reported outcomes that is completed weekly on a mobile application device used clinically to track spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis
* To be listed for lung transplant
* Has purchased home spirometer

Exclusion Criteria:

* Diagnosis other than Cystic Fibrosis
* Unable to read
* Unable to use computer or smartphone device to access mobile application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Lung Allocation Score (LAS) | Through study completion, an average of 3-6 months (time spent on the lung transplant waiting list).
  Change in LAS value at the first clinic visit triggered by the clinical tool

SECONDARY OUTCOMES:
Time to transplant | Through study completion, up to 1 year
  Measured in days (time spent on the lung transplant waiting list)
Survival to transplant | Through study completion, up to 1 year
  Binary outcome measure to indicate if individual survived to transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No